CLINICAL TRIAL: NCT01403844
Title: Skin Carotenoid Response to Intake of Vegetables and Fruits Recommended by the Dietary Guidelines
Brief Title: Carotenoid Response to the Intake of Vegetables and Fruits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GFHNRC022
Record Dates: First submitted 2011-07-21; First posted 2011-07-27 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Resonance Raman Spectroscopy for Dietary Carotenoid Intake
Keywords: resonance Raman spectroscopy; Dietary Guidelines; fruits; biomarkers; carotenoids; MyPlate; vegetables

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Skin Carotenoids (Other): Skin carotenoids will be measured under conditions of depletion or repletion
  Interventions: Other: Carotenoid Depletion; Other: Carotenoid Repletion; Other: Natural Repletion

INTERVENTIONS:
Other: Carotenoid Depletion — Depletion of carotenoids using a restricted food list
Other: Carotenoid Repletion — Carotenoid repletion with provided diet based on dietary guidelines.
Other: Carotenoid Depletion — Carotenoid depletion using a restricted food list.
Other: Natural Repletion — Resumption of usual personal diet regimen. No restrictions.

SUMMARY:
The purpose of this study is to validate the non-invasive tool, resonance Raman spectroscopy for assessing vegetable and fruit consumption.

DETAILED DESCRIPTION:
This study will validate the use of resonance Raman spectroscopy to assess vegetable and fruit intake by performing a controlled feeding study during which volunteers will consume a provided diet with known amounts of carotenoids in the form of fruits and vegetables.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 - 65 years
* Weight stable (±5 lbs) for at least 2 months prior to the start of the study
* Body mass index (BMI) between 19-30 kg/m2
* Willing to refrain from the use of nicotine and dietary supplements for the duration of the study
* Willing to maintain baseline weight and physical activity levels

Exclusion Criteria:

1. BMI greater than 30.
2. Gastrointestinal disorders, disease, or medication that affects carotenoid absorption or storage
3. Current smoker
4. Allergies or intolerances to foods to be utilized in the study
5. Consumption of greater than an average of 1 alcoholic drink/day for women and 2/day for men, use of nutritional/sports supplements (if unwilling to discontinue during the study)
6. Pregnancy or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Serum and skin levels of carotenoids in adults fed a high carotenoid diet | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James Roemmich, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jahns L, Johnson LK, Mayne ST, Cartmel B, Picklo MJ Sr, Ermakov IV, Gellermann W, Whigham LD. Skin and plasma carotenoid response to a provided intervention diet high in vegetables and fruit: uptake and depletion kinetics. Am J Clin Nutr. 2014 Sep;100(3):930-7. doi: 10.3945/ajcn.114.086900. Epub 2014 Jul 9. PMID 25008856
- See also: Grand Forks Human Nutrition Research Center — https://www.ars.usda.gov/plains-area/gfnd/gfhnrc/